CLINICAL TRIAL: NCT00090337
Title: Acupuncture for Pain and Dysfunction Following Neck Dissection: A Randomized, Controlled, Phase III Trial
Brief Title: Acupuncture or Standard Therapy in Treating Pain and Dysfunction in Patients Who Have Undergone Neck Surgery for Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: David G. Pfister, Memorial Sloan-Kettering Cancer Center
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: 03-131; R21CA098792 (NIH); P30CA008748 (NIH); MSKCC-03131A
Record Dates: First submitted 2004-08-25; First posted 2004-08-26 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer; Pain
Keywords: pain; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms | interventions — Acupuncture Therapy

ARMS (2):
- Arm I (Experimental): Patients undergo acupuncture for 20-30 minutes once weekly for 4 weeks.
  Interventions: Procedure: acupuncture therapy
- Arm II (Active Comparator): Patients undergo standard of care for 4 weeks.
  Interventions: Procedure: standard follow-up care

INTERVENTIONS:
Procedure: acupuncture therapy — Patients undergo acupuncture for 20-30 minutes once weekly for 4 weeks
  Arms: Arm I
Procedure: standard follow-up care — Patients undergo standard care
  Arms: Arm II

SUMMARY:
RATIONALE: Acupuncture may help relieve pain and dysfunction caused by cancer surgery. It is not yet known whether acupuncture is more effective than standard therapy in treating pain and dysfunction in patients who have undergone neck surgery for head and neck cancer.

PURPOSE: This randomized phase III trial is studying acupuncture to see how well it works compared to standard therapy in treating pain and dysfunction in patients who have undergone neck surgery for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether acupuncture reduces pain and dysfunction in patients with head and neck cancer who have undergone neck dissection.

Secondary

* Determine whether acupuncture relieves dry mouth in these patients.

OUTLINE: This is a randomized, controlled study. Patients are stratified according to surgical procedure (selective neck dissection vs modified radical neck dissection vs radical neck dissection) and baseline Constant-Murley score (≤ 35 vs > 35). Patients are randomized into 1 of 2 treatment arms.

* Arm I: Patients undergo acupuncture for 20-30 minutes once weekly for 4 weeks.
* Arm II: Patients undergo standard of care for 4 weeks. In both arms, treatment continues in the absence of unacceptable toxicity.

The Constant-Murley score is assessed at baseline and then at week 6. Pain medication use is recorded at baseline, during study treatment, and then at week 6. Numerical Rating Scale of pain on activity and xerostomia inventories are completed at baseline and then at weeks 5 and 6.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 58 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must have undergone neck dissection for cancer ≥ 3 months ago (in order to qualify pain as chronic sequella)
* Subjective complaint of pain and/or dysfunction in the neck and/or shoulders that, in the opinion of the investigator, is due to neck dissection
* Constant-Murley score ≤ 70 (i.e., moderate or severe pain and dysfunction)
* No moderate or severe neck or shoulder pain that, in the opinion of the investigator, is not due to cancer surgery

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 months since prior radiotherapy
* More than 6 weeks since prior acupuncture
* Concurrent analgesics allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2003-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pain, function and activities of daily living as measured by the Constant-Murley instrument

SECONDARY OUTCOMES:
Xerostomia as measured by the Xerostomia Inventory questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David G. Pfister, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan - Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Result] Pfister DG, Cassileth BR, Deng GE, Yeung KS, Lee JS, Garrity D, Cronin A, Lee N, Kraus D, Shaha AR, Shah J, Vickers AJ. Acupuncture for pain and dysfunction after neck dissection: results of a randomized controlled trial. J Clin Oncol. 2010 May 20;28(15):2565-70. doi: 10.1200/JCO.2009.26.9860. Epub 2010 Apr 20. PMID 20406930